CLINICAL TRIAL: NCT00595699
Title: Escitalopram Treatment of Major Depression in Patients With Temporal Lobe Epilepsy. A Double-blind, Placebo-controlled Study.
Brief Title: Escitalopram Treatment of Major Depression in Patients With Temporal Lobe Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Conrad, Erich J., M.D. (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Erich J. Conrad, M.D., LSUHSC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LXP-MD-116; LSUHSC IRB #6653
Record Dates: First submitted 2008-01-03; First posted 2008-01-16 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2008-01

CONDITIONS: Major Depression; Temporal Lobe Epilepsy
MeSH Terms: conditions — Depressive Disorder, Major; Epilepsy, Temporal Lobe | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Double-blind
  Interventions: Drug: placebo
- 1 (Experimental): escitalopram group
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram — 10 mg daily for the first week followed by an increase to 20 mg daily for the remainder of the study
  Other Names: Lexapro
  Arms: 1
Drug: placebo — Placebo
  Arms: 2

SUMMARY:
This is a research study evaluating the use of escitalopram (Lexapro®) for the treatment of major depression in subjects with temporal lobe epilepsy. The purpose of the study is to measure the severity and change in depressive and anxiety symptoms after 10 weeks of study treatment with escitalopram or placebo as measured by certain rating scales and questionnaires. In addition, the study will measure the frequency of seizures using a patient diary during the study. Finally, the study will assess the change in the quality of life using rating scales.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a confirmed diagnosis of temporal lobe epilepsy
2. Subject meets DSM-IV criteria for Major Depression
3. MADRS greater than or equal to 15 at screening and baseline
4. Subject between ages of 18 and 65
5. Female subjects of childbearing potential must take adequate contraceptive precautions (methods with a published failure rate of less than 1% per year, or condom/diaphragm, or diaphragm/spermicide)
6. Subject must provide voluntary signed informed consent approved by the Institutional Review Board of LSU Health Sciences Center

Exclusion Criteria:

1. Any other primary axis I diagnosis other than Major Depression
2. The presence of psychogenic, non-epileptic seizures
3. A history of non-response to two or more antidepressants given for an adequate therapeutic trial
4. The presence of substance abuse or dependence in past six months
5. The presence of clinically significant malnutrition, cardiac, hepatic or renal disease that might endanger the safety of the subject
6. Pregnancy or nursing
7. Any subjects with suspected mental retardation, psychotic disorder or dementia
8. Subjects whose anticonvulsant medication regimen includes phenobarbital
9. Individuals who will require psychotropic medications such as benzodiazepines or medications likely to cause significant effects on mood or anxiety as outlined in section 5.4
10. Cognitive-behavioral therapy will not be allowed during the course of the study. Other psychotherapeutic modalities (supportive, psychoanalytic, etc.) will be allowed only if the individual has been in therapy for the previous 12 weeks and plans to remain in therapy throughout the duration of the study.
11. Individuals who in the opinion of the investigator would not be able to understand or comply with study requirements
12. Individuals with a known hypersensitivity to escitalopram or any of its ingredients
13. Individuals who in the opinion of the investigator present a significant risk of suicide, or have had a significant suicide attempt in the past two years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Montgomery And Asberg Depression Rating Scale | Screen, Baseline, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 10

SECONDARY OUTCOMES:
Clinician's Global Impression Severity and Improvement subscales | Baseline, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Erich J Conrad, M.D, Principal Investigator — LSUHSC
Locations (1):
- LSU Anxiety and Mood Disorders Clinic, New Orleans, Louisiana, United States